CLINICAL TRIAL: NCT04077203
Title: Biofeedback of Glucose in Non-diabetic Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klick Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00036792
Record Dates: First submitted 2019-08-29; First posted 2019-09-04 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2019-09

CONDITIONS: Blood Glucose; Biofeedback
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Sham Comparator): Those receiving no visual feedback because the handheld device monitor will be occluded with black tape (the control group).
  Interventions: Behavioral: Biofeedback / No biofeedback
- Test (Experimental): Those receiving the ability to visualize their glucose levels via the handheld device (the biofeedback group).
  Interventions: Behavioral: Biofeedback / No biofeedback

INTERVENTIONS:
Behavioral: Biofeedback / No biofeedback — Biofeedback / No biofeedback

SUMMARY:
This research examines whether biofeedback of glucose (i.e., knowledge of one's own glucose levels) in non-diabetic participants affects their health behaviours (e.g., eating, nutrition, exercise, etc.). This study utilizes wearable continuous glucose (CGM) technology, which provides personalized feedback to participants to allow them to self-monitor their own glucose levels.

DETAILED DESCRIPTION:
The purpose of this research is to examine whether self-monitoring and biofeedback of glucose levels improves health outcomes in non-diabetic participants. All participants will receive a continuous flash glucose monitor (consisting of an adhesive patch sensor and a handheld reader device) to wear for 14 days. Participants will be randomized into one of 2 groups: those receiving biofeedback (the ability to visualize their glucose levels via the handheld device), and the control group (receiving no biofeedback because the handheld device monitor will be occluded with black tape). Participants' objective and self-report health metrics will be measured before and after the 14-day intervention. The goal is to examine whether the biofeedback condition influences any daily activities or physiological measurements compared to the control condition, as a direct result of self-monitoring glucose levels.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Below the age of 18 years
* Diagnosis of any known chronic or acute medical disease (e.g., diabetes, cardiovascular disease, respiratory disease, influenza, pneumonia, etc.)
* Diagnosis of any known neurological disease or psychological disorder (e.g., brain lesion, epilepsy, anxiety, eating disorder, mood disorder, sleep disorder, etc.)
* Any implanted electrical medical device (e.g., pacemaker, insulin pump, deep brain stimulator, etc.)
* Suspected or confirmed pregnancy
* Currently breastfeeding
* Use of antibiotics in the three months prior to enrollment
* Any person planning to undergo a Magnetic Resonance Imaging (MRI), Computed Tomography (CT) scan, or high-frequency electrical heat (diathermy) treatment during the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Weight in kg | 2 weeks
  Weight in kg
Body Mass Index (BMI) | 2 weeks
  Height in cm and weight in kg will be used to calculate BMI
Body fat % | 2 weeks
  Using a smart scale
Resting heart rate | 2 weeks
  Using a sphygmomanometer with heart rate sensor
Resting blood pressure (systolic and diastolic) | 2 weeks
  Using a sphygmomanometer
Self-reported positive and negative affect | 2 weeks
  Positive and Negative Affect Schedule (PANAS; Watson et al., 1988). The scale consists of 20 items (10 for Positive Affect; 10 for Negative Affect), with each item rated on a 5-point scale of 1 (not at all) to 5 (extremely). Items are summed for Positive affect and Negative affect, with higher scores indicating a higher level of affect in each respective scale.
Self-reported general health | 2 weeks
  12-Item Short-Form Health Survey (SF-12; Ware et al., 1996). The scale measures overall general self-reported physical and mental health using 12 items, on 2 to 6-point ordinal scales. The range of possible total scores is 12 to 48, with higher scores indicating better health.
Self-reported perceived stress | 2 weeks
  Perceived Stress Scale (Cohen et al., 1983; Cohen & Williamson, 1988). This is a 4-item scale that measures overall stress with each item evaluated on a 5-point Likert scale. The range of possible total scores is 0 to 16, with higher scores indicating more stress.
Self-reported sleep quality | 2 weeks
  Pittsburgh Sleep Quality Index (Buysse et al., 1989). This is a 19-item scale that measures self-reported sleep quality and sleep disturbances, comprised of open-ended questions and scaled items evaluated on a 4-point Likert scale. The range of possible total scores is 0 to 21, with higher scores indicating poorer sleep quality.
Self-reported general well-being | 2 weeks
  Satisfaction with Life Scale (Diener et al., 1985). This is a 5-item scale that measures overall well-being with each item evaluated on a 7-point Likert scale. The range of possible total scores is 5 to 35, with higher scores indicating higher well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Klick Inc., Toronto, Ontario, Canada